CLINICAL TRIAL: NCT04637906
Title: Short and Long-term Effects of Adding Oral L-arginine to Standard Therapy in Patients With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Randomized, Parallel Group, Double-blind Placebo-controlled Clinical Trial
Brief Title: Short and Long-term Effects of Adding Oral L-arginine to Standard Therapy in Patients With COVID-19 (SARS-CoV-2)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, giuseppe fiorentino, PROFESSOR, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Bioarginina
Record Dates: First submitted 2020-11-18; First posted 2020-11-20 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-arginine (Experimental): Bioarginina®, 2 orally administered vials per day
  Interventions: Dietary Supplement: Bioarginina®
- Placebo (Placebo Comparator): 2 orally administered vials per day of Bioarginina® without L-arginine
  Interventions: Dietary Supplement: Bioarginina®

INTERVENTIONS:
Dietary Supplement: Bioarginina® — Food supplement based on 1,66 grams of L-arginine

SUMMARY:
Single-center study with a parallel group scheme, double-blind, randomized, placebo-controlled, to evaluate whether the addition to the investigator's hospital standard therapy of two vials of Bioarginina® per day in subjects with SARS-CoV-2 is useful for treatment of this pathology.

DETAILED DESCRIPTION:
Preliminary experiences conducted in patients affected by SARS-CoV-2 infection by adding the daily oral administration of two vials of Bioarginina® to the standard therapy have shown favorable effects on discharge times, on the recovery of the number of lymphocytes and on the P \ F ratio between arterial pO2 and FiO2 breathed. In particular, for the latter parameter there is almost a doubling of the recovery speed.

The investigators therefore, decided to undertake the present spontaneous, single-center study with a parallel group scheme, double-blind randomized, placebo-controlled to evaluate whether the addition to the standard therapy of two vials per day of Bioarginina® in subjects of our hospital suffering from SARS-CoV-2 is useful for the treatment of this pathology.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* Diagnosis of COVID 19, confirmed by RT-PCR on a nasopharyngeal swab
* COVID 19 pneumonia with the following clinical characteristics: SpO2 in ambient air <93% and Alveolar pressure of oxygen / inspiratory fraction of oxygen (PaO2 / FiO2 - P / F <300 mmHg.
* Lymphocytopenia defined as lymphocytes <1500 / mcL or <20% of white blood cells

Exclusion Criteria:

* History of intolerance to L-arginine
* Severe chronic pulmonary disease
* Pregnancy or breastfeeding
* Neutropenia due to neoplasms of the haematopoietic system or other organs with invasion of the bone marrow
* Use of immunosuppressive drugs or cytotoxic chemotherapies within the previous three weeks
* Refusal to give consent to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-04-18 (Estimated); Study Completion 2021-09-18 (Estimated)

PRIMARY OUTCOMES:
Reduction of P / F normalization times | 60 days
  Alveolar pressure of oxygen / inspiratory fraction of oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Fiorentino, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Azienda Ospedaliera Specialistica Dei Colli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fiorentino G, Coppola A, Izzo R, Annunziata A, Bernardo M, Lombardi A, Trimarco V, Santulli G, Trimarco B. Effects of adding L-arginine orally to standard therapy in patients with COVID-19: A randomized, double-blind, placebo-controlled, parallel-group trial. Results of the first interim analysis. EClinicalMedicine. 2021 Oct;40:101125. doi: 10.1016/j.eclinm.2021.101125. Epub 2021 Sep 9. PMID 34522871